CLINICAL TRIAL: NCT02670824
Title: Study to Determine the Safety, Tolerability, and Pharmacokinetics of a Single Escalating Dose and Repeated Doses of CN-105 in Healthy Adult Subjects
Brief Title: Safety Study of CN-105 Neuroprotective Peptide for Intracerebral Hemorrhage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AegisCN LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN-105-01
Record Dates: First submitted 2016-01-07; First posted 2016-02-02 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Intracerebral Hemorrhage (ICH)
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — apolipoprotein E mimetic peptide CN-105

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CN-105 Active Drug (Experimental): The CN-105 drug administered via IV at an escalating scale of mg/kg.
  A1-0.01 mg/kg A2-0.03 mg/kg A3-0.1 mg/kg A4-0.3 mg/kg A5-1.0 mg/kg B1-1.0 mg/kg
  Interventions: Drug: CN-105
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CN-105 — Single and multiple intravenous (IV) doses of CN-105
  Arms: CN-105 Active Drug
Drug: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
This study evaluates the safety, tolerability, and pharmacokinetics (PK) of a single escalating dose and repeated doses of CN-105 in healthy adult participants. There will be about 48 subjects, 36 active and 12 placebo.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH), which is often associated with longstanding hypertension, affects as many as 50,000 people annually in the United States alone. ICH remains associated with poor outcome, and approximately 40 to 50% of afflicted patients will die within 30 days. Unfortunately, little improvement has been made in the ICH-associated mortality rate over the last 20 years. To address this issue, the National Institutes of Health issued a priorities report in 2005, and the American Heart Association released a recent set of clinical guidelines for the first time in nearly a decade. In these reports, the importance of developing clinically relevant models of ICH that will extend our understanding of the pathophysiology of the disease and target new therapeutic approaches was emphasized. At present, however, there are no proven neuroprotective pharmacological treatments for ICH or other forms of acute brain injuries, such as traumatic brain injury (TBI) and subarachnoid hemorrhage (SAH).

To meet this unmet medical need, CereNova, LLC has developed a novel therapeutic approach based on the known biological function of endogenous apolipoprotein E (apoE), a key mediator of the neuroinflammatory response and recovery from a variety of acute and chronic brain injuries1-5. There are three common human isoforms of apolipoprotein E, designated apoE2, apoE3, and apoE4, which differ by single cysteine to arginine substitutions at positions 112 and 158. Although originally defined in the context of cholesterol metabolism, apoE is also produced in the brain, where it modulates neuroinflammatory responses and functional outcomes after injury in an isoform specific fashion1. Specifically, the apoE3 protein isoform plays an adaptive role in downregulating glial activation and reducing secondary neuronal injury, whereas the E4 isoform is associated with increased neuroinflammation and poor functional outcomes.

Although the intact apoE holoprotein does not cross the blood brain barrier (BBB) and thus cannot be administered therapeutically, we have previously demonstrated that smaller apoE mimetic peptides do effectively cross the BBB while effectively downregulating the brain inflammatory responses in vitro and in vivo6. CN-105, CereNova's lead clinical candidate, is a small, 5 amino acid apoE-mimetic peptide that is derived from the receptor binding region of apoE. CN-105 retains the anti-inflammatory and neuroprotective effects of intact apoE, is well tolerated in preclinical studies, and readily crosses the BBB to effectively reduce inflammatory responses in the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written Informed Consent to participate in the study prior to undergoing any screening procedures.
2. Non-smoking and does not use nicotine-containing products (including smoking cessation aids, such as gums or patches) for 6 months or greater at study commencement
3. Adult male or female volunteers between 18 and 50 years (inclusive) at screening
4. BMI between 18-33 kg/m2 (inclusive) and weighing at least 110 lbs (50 kg).
5. Healthy on the basis of the medical history, physical examination, vital signs, ECG, blood chemistry, hematology, and urinalysis performed at screening.
6. Adequate peripheral forearm vein access.
7. No significant dietary restrictions and willing to fully consume all Duke CRU "Regular Diet" meals and beverages/water provided to them.
8. No prescription medication except contraception as described in Inclusion #10 within 7 days or 5 half-lives (whichever is longer) of study entry (randomization and initiation of study drug administration) or any over-the-counter (OTC) medication or herbal/vitamin supplement within 7 days of study entry, and not expected to require or take any prescription or over-the-counter medication or supplement for the full duration of the study. Acetaminophen at doses of ≤1 g/day may be used and stable treatment for seasonal allergies (other than glucocorticoids via any route) may be used. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
9. Women who are of non-childbearing potential, must be:

   Surgically sterile (removal of both ovaries and/ or uterus at least 12 months prior to dosing).

   Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing on Day -1 and with an FSH level at screening of ≥ 40 mIU/mL.
10. Women of child-bearing potential must have a negative serum pregnancy test at screening and urine pregnancy test during the study, and must agree to avoid pregnancy during study and for three months after the last dose of study drug. Pregnancy is tested at screening, during check-in, during the follow-up visit, and at any given point if deemed necessary to the PI or designate. During treatment, women of child-bearing potential must use two acceptable methods of contraception at the same time unless the subject has had a documented tubal sterilization or chooses to use a Copper T 380A IUD or LNG 20 IUS, in which case no additional contraception is required. Medically acceptable contraceptives include: (1) documented surgical sterilization (such as a hysterectomy), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, (3) hormonal contraception (combination oral contraceptives, transdermal patch, injectables, implantables, or vaginal ring) or (4) an intrauterine device (IUD) or intrauterine system (IUS). Abstinence is not an acceptable form of contraception in this study.
11. Male participants must agree to take all necessary measures to avoid causing pregnancy in their sexual partners during the study and for three months after the last dose of study drug. Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicidal. Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use.
12. Must not have donated blood, platelets, or any other blood components 30 days, or plasma 90 days, prior to consenting. Must also agree not to donate blood, platelets, or any other blood components for 3 months after the last dose of study drug.
13. Male participants must agree not to donate sperm during the study and for 12 weeks after the last dose.
14. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Laboratory results outside the normal range, if considered clinically significant (CS) by the PI or delegate. Any laboratory result outside the normal range and not clinically significant will be designated as such by NCS (Non-clinically Significant).
2. Mental capacity that is limited to the extent that the participant cannot provide legal consent or understand information regarding the side effects of the study drug.
3. Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years or drinks more than 3 cups of coffee per day.
4. Unwillingness or lack of ability to comply with the protocol, or to cooperate fully with the PI and site personnel.
5. Clinically significant ECG abnormality in the opinion of the PI or delegate.
6. Has taken any other investigational drug during the 30 days or 5 half-lives (whichever is longer) prior to the screening visit or is currently participating in another investigational drug clinical trial.
7. History or manifestation of clinically significant neurological (e.g., frequent headaches or migraines), gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematologic or other medical disorders that might influence the interpretation of the results of the study.
8. Infected with Hepatitis B or C or HIV Virus.
9. Participants who have a history of unexplained syncope or fainting from the collection of blood; i.e., autonomic dysfunction.
10. Lack of ability to understand verbal and/ or written English
11. Subjects who had significant trauma or surgical procedure within 1 month prior to Screening.
12. A positive urine drug screen or positive alcohol breathalyzer test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The number and percentage of participants having study procedure-related suspected adverse reactions assessed by change from baseline in vital signs, ECG and clinical labs. | up to 1 week
  The number and percentage of participants having study procedure-related suspected adverse reactions assessed by change from baseline in vital signs, ECG and clinical labs will be tabulated and evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Wangqin R, Meng X, Li H, Wang Y, Wang H, Laskowitz D, Chen X, Wang Y. Tolerability and Pharmacokinetics of Single Escalating and Repeated Doses of CN-105 in Healthy Participants. Clin Ther. 2022 May;44(5):744-754. doi: 10.1016/j.clinthera.2022.03.006. Epub 2022 May 11. PMID 35562205